CLINICAL TRIAL: NCT01683721
Title: The UNMASK Study: A Post-Market Longitudinal Observational Study of the WinxTM Sleep Therapy System for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: Post-Market Observational Study of the WINX Sleep Therapy for the Treatment of Obstructive Sleep Apnea (OSA)
Acronym: UNMASK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ApniCure, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12023
Record Dates: First submitted 2012-09-07; First posted 2012-09-12 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Winx

SUMMARY:
The objective of the Study is to observe the use and utility of the Winx Sleep Therapy System in a clinical practice, for the treatment of patients with obstructive sleep apnea (OSA).

ELIGIBILITY:
Exclusion Criteria

* Has a severe respiratory disorder, such as severe lung disease, pneumothorax, etc.
* Has loose teeth or advanced periodontal disease.
* Is under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with obstructive sleep apnea (OSA)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - St. Petersburg Sleep Disorders Center, St. Petersburg, Florida
  - Sleep Medicine Associates of Texas (SMAT), Dallas, Texas